CLINICAL TRIAL: NCT00404300
Title: An Open Multi-centre Study to Investigate the Safety and Efficacy of OPTIVATE®, a High Purity, Dual Inactivated Factor VIII and Von Willebrand Factor Concentrate, in Patients With Von Willebrand Disease Who Are Undergoing Surgery
Brief Title: Optivate in People With Von Willebrand Disease Undergoing Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow recruitment and a delay in reaching the recruitment target.
Sponsor: Bio Products Laboratory (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8VWF03
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — optivate

INTERVENTIONS:
Drug: Optivate — Plasma-derived Factor VIII

SUMMARY:
An open, multi-centre study in patients with von Willebrand Disease (VWD) undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent.
2. Be aged 12 years or older.
3. Have VWD of known type.
4. Be due to undergo surgery, in which the investigator believes a VWF concentrate will be required.
5. Have a known lack of, poor response to, or contraindication to, DDAVP, or require a type of surgery in which a plasma-derived product is appropriate.
6. Have a prothrombin time (PT) of not more than 3 seconds above the upper limit of the reference range.
7. Female patients of child-bearing potential, with the exception of pregnant patients undergoing Caesarean surgery or other modes of delivery, including normal vaginal delivery, must have a negative result on a human chorionic gonadotropin-based pregnancy test. If a female patient is or becomes sexually active, she must practice contraception by using a method of proven reliability for the duration of the study.

Exclusion Criteria:

1. Have a history of inhibitor development to VWF or FVIII or a positive result at screening (positive screen for VWF inhibitor; positive screen and a result of >0.5 BU for FVIII inhibitor). A result at screening is not mandatory if the patient is to undergo emergency surgery and the local laboratory is unable to perform the analyses.
2. Patients with thrombocytopenia (platelets <50 x 109/L).
3. Patients who have clinically significant renal disease (creatinine >200 µmol/L).
4. Patients who have clinically significant liver disease (ALT levels greater than three times the upper limit of the reference range).
5. Presence of any other major systemic illnesses which would compromise the outcome of the study in the opinion of the investigator.
6. Known or suspected hypersensitivity to investigational medicinal product (IMP) or its excipients.
7. Have a recent history of alcohol or drug abuse.
8. Administration of a new chemical entity within the 4 months preceding enrolment.
9. Participation in any other clinical study in which investigational or marketed drugs were employed in the 30 days preceding enrolment (screening visit) into this study, with the exception of the BPL clinical study Protocol 8VWF01.
10. Female patients who are lactating.
11. In the opinion of the investigator, the patient is unlikely to comply with the study protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-02; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
A subjective overall assessment by the investigator of OPTIVATE® in the control of bleeding due to surgery throughout the whole study. | Throughout the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Thynn Thynn Yee, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (4):
- Israel (3):
  - Rambam Health Care Campus, 8 Haaliya St., Bat-Galim, Haifa
  - Haddasah Ein-Karem Medical Center, P.O.Box 12000, Jerusalem
  - Beilinson Hospital, Rabin Medical Center, 39 Jabotinsky Street, Petah Tikva
- Katharine Dormandy Haemophilia Centre and Haemostasis Unit, Royal Free Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor's homepage — http://www.bpl.co.uk